CLINICAL TRIAL: NCT03880877
Title: Regorafenib Plus FOLFIRI With Irinotecan Dose Escalated According to UGT1A1 Genotyping Versus Regorafenib Monotherapy in Patients With Previously Treated Metastatic Colorectal Cancer: A Prospective, Randomized, Controlled Study
Brief Title: Regorafenib Plus FOLFIRI With Irinotecan Dose Escalated in Patients With Previously Treated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Vice Superintendent, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20190032
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; FOLFIRI; regorafenib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib plus FOLFIRI (Experimental): Regimen for treatment consists of irinotecan (180 mg/m2 as a 120-min IV infusion for UGT1A1 genotyping (TA6/TA6) and UGT1A1 genotyping (TA6/TA7); 120 mg/m2 as a 120-min IV infusion for UGT1A1 genotyping (TA7/TA7)), followed by Leucovorin (400 mg/m2 IV infusion over 2 hours), and fluorouracil (5-FU) (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  After every 2 cycles of each different dose of irinotecan, if adverse events (AEs) are under the grade 2, we will escalate the dose of 30 mg/m2. The estimated maximal dose of irinotecan is 260 mg/m2 for UGT1A1 genotyping (TA6/TA6); 240 mg/m2 for UGT1A1 genotyping (TA6/TA7); 180 mg/m2 for UGT1A1 genotyping (TA7/TA7).
  Regorafenib is administered at adjusted dosage of 120 mg daily for 3 weeks in a 4-week cycle.
  Interventions: Drug: Regorafenib; Genetic: UGT1A1 genotyping (TA6/TA6); Genetic: UGT1A1 genotyping (TA6/TA7); Genetic: UGT1A1 genotyping (TA7/TA7); Drug: Leucovorin and 5-FU
- Regorafenib (Active Comparator): Regorafenib is administered at adjusted dosage of 120 mg daily for 3 weeks in a 4-week cycle.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is administered at dose of 120 mg daily for 3 weeks in a 4-week cycle
  Other Names: stivarga
Genetic: UGT1A1 genotyping (TA6/TA6) — The dosage of irinotecan in FOLFIRI is escalated from 180mg/m2 to 260 mg/m2
  Arms: Regorafenib plus FOLFIRI
Genetic: UGT1A1 genotyping (TA6/TA7) — The dosage of irinotecan in FOLFIRI is escalated from 180mg/m2 to 240 mg/m2
  Arms: Regorafenib plus FOLFIRI
Genetic: UGT1A1 genotyping (TA7/TA7) — The dosage of irinotecan in FOLFIRI is escalated from 120mg/m2 to180 mg/m2
  Arms: Regorafenib plus FOLFIRI
Drug: Leucovorin and 5-FU — Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period)
  Arms: Regorafenib plus FOLFIRI

SUMMARY:
A prospective, multicenter, randomized in a 2:1 ratio, controlled, clinical trial with two parallel arms will be conducted to compare irinotecan dose escalated FOLFIRI according to UGT1A1 genotyping plus 120 mg regorafenib with 120 mg regorafenib alone in previously treated patients with metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Primary objective:

Progression-free survival

Secondary objective:

Overall survival, best objective response, disease control rate, time to progression, duration of treatment and adverse events

Number of Subjects: 153 patients with metastatic colorectal cancer treated with regorafenib and FOLFIRI as a third- or fourth-line setting.

Plan of the Study:

1. This is a prospective, multicenter, randomized in a 2:1 ratio, controlled study.
2. Study Schedule Study date: the time getting approval letter issued by both regulatory authority and institutional review board (IRB). Duration of the study: 4 years.
3. Duration of Treatment: Treatment was administered until disease progressed.

ELIGIBILITY:
Inclusion Criteria:

1. Cyto-/histological confirmed mCRC
2. Patients who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib as 3rd line (RAS mutant) or 4th line (RAS wild type) therapy
3. Aged no less than 20 years, at the time of acquisition of informed consent
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
5. Patients with measurable or non-measurable disease in the colon or rectum, according to RECIST criteria version 1.1
6. Life expectancy more than 12 weeks
7. Women with childbearing potential must agree to perform adequate contraception measures since informed consent till a least 12 weeks after the last study drug administration.

   The investigators or designee are requested to advise the patient to achieve adequate birth control.
8. Adequate organ and bone marrow function as defined below:

   * Total bilirubin <= 1.5 x the upper limit of normal (ULN)
   * Alanine amino-transferase (ALT) and aspartate amino-transferase (AST) <= 2.5 x ULN (<= 5 x ULN for patients with liver metastases)
   * Alkaline phosphatase (ALP) <= 2.5 x ULN (<= 5 x ULN for patients with liver metastases)
   * Amylase and lipase <= 1.5 x ULN
   * Serum creatinine <= 1.5 x ULN
   * Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m2, according to the modified diet in renal disease (MDRD) abbreviated formula
   * International normalized ratio (INR)/partial thromboplastin time (PTT) <= 1.5 x ULN
   * Platelet counts >= 100,000/mm3
   * Hemoglobin level >= 9 g/dL
   * Absolute neutrophil counts >= 1,500/mm3
9. Ability to understand and willingness to sign written Informed Consent Form (ICF)

Exclusion Criteria:

1. Prior treatment with regorafenib within 28 days
2. Other concurrent cancer or prior treatment for other carcinomas within the last five years, except curatively treated non-melanoma skin cancer, superficial bladder tumors, and cervical cancer in-situ
3. Extended field radiotherapy within 28 days or limited radiotherapy within 14 days prior to randomization
4. Major surgery within 28 days prior to start of study treatment (diagnostic biopsy, laparotomy, line placement is not considered as major surgery)
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction in the past 12 months, active gastrointestinal bleeding, central nervous system disorders or psychiatric illness/social situation that would limit compliance with study requirements or judged to be ineligible for the study by the investigator
6. History of myocardial infarction, deep venous or arterial thrombosis, or cardiovascular accident (CVA) during the last 6 months
7. Uncontrolled cardiac arrhythmias, unstable angina, or newly-onset angina within 3 months prior to study entry
8. Uncontrolled hypertension despite optimal management (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg)
9. Patients with known central nervous system (CNS) metastases
10. Having received any investigational agents or participating in any investigational drug study within 4 weeks prior to study enrollment
11. Pregnant or breast-feeding female (a pregnancy test must be performed on all female patients with child-bearing potential within 7 days of treatment initiation, and the result must be negative)
12. Inability to take oral medications
13. Poor compliance as judged by the investigator

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of initiation of treatment until the date of first documented progression, assessed up to 23 months
  Time from treatment to disease progresses and lives

SECONDARY OUTCOMES:
Overall survival | From date of initiation of treatment until the date of death from any cause, assessed up to 23 months
  Time from treatment to death of patients
Best objective response | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  best response recorded during treatment
Disease control rate | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  Rate of best objective response, including complete response, partial response and stable disease
Time to progression | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  Time from treatment to disease progresses
Duration of treatment | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  Time from initiation to termination of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, PhD, Study Chair — Division of Colorectal Surgery, Department of Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CW, Chen YC, Ker TW, Lin YW, Chang TK, Su WC, Chen PJ, Tsai HL, Wang JY. Efficacy and safety of regorafenib plus FOLFIRI with UGT1A1 genotyping-guided irinotecan dose escalation against metastatic colorectal cancer: a multicenter, phase II, open-label, two-arm randomized controlled tria. Ther Adv Med Oncol. 2025 Oct 23;17:17588359251371489. doi: 10.1177/17588359251371489. eCollection 2025. PMID 41164204
- [Derived] Ma CJ, Chang TK, Tsai HL, Su WC, Huang CW, Yeh YS, Chang YT, Wang JY. Regorafenib plus FOLFIRI with irinotecan dose escalated according to uridine diphosphate glucuronosyltransferase 1A1genotyping in previous treated metastatic colorectal cancer patients:study protocol for a randomized controlled trial. Trials. 2019 Dec 19;20(1):751. doi: 10.1186/s13063-019-3917-z. PMID 31856912